CLINICAL TRIAL: NCT07351162
Title: Hypertension Treatment in Nigeria Program 2.0
Brief Title: Hypertension Treatment in Nigeria 2.0
Acronym: HTN 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Abuja Teaching Hospital (Other); University of Abuja (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mark Huffman, William Bowen Professor of Medicine, Professor of Public Health, Co-Director Global Health Center and Global Health Futures, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UATH/HREC/PR/557/A2; R01HL144708 (NIH)
Record Dates: First submitted 2026-01-15; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hypertension (HTN)
Keywords: Hypertension; Nigeria; Primary Health Center; HEARTS technical package
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This study applies an interrupted time series design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Health Care Centers (Experimental): 50 primary healthcare centers across five Nigerian states will be selected to implement a hypertension treatment program based on the WHO HEARTS hypertension technical package.
  Interventions: Other: Implementation of a modified WHO HEARTS Hypertension Treatment Bundle

INTERVENTIONS:
Other: Implementation of a modified WHO HEARTS Hypertension Treatment Bundle — The intervention seeks to the scale-up of the World Health Organization HEARTS package in 50 primary healthcare centers across five Nigerian states using a type II hybrid effectiveness implementation design. Following a 12-month pre-implementation period, centers will transition into a 24-month implementation period that includes state-level training of health workers, non-physician hypertension screening, diagnosis, and treatment, simplified hypertension treatment guidelines, monthly audit and feedback, supply chain strengthening, and a drug revolving fund to improve blood pressure lowering medication accessibility.

SUMMARY:
The purpose of the second phase of the Hypertension Treatment in Nigeria (HTN 2.0) Program is to build upon the success of the first phase of the HTN Program (2020-2023), which implemented the WHO HEARTS package across 60 primary healthcare centers (PHCs) in the Federal Capital Territory, Nigeria. This program demonstrated significant improvements in hypertension treatment and control. HTN 2.0 will expand implementation of the HEARTS bundle to 5 new states in 5 geopolitical zones in Nigeria (Abia, Delta, Gombe, Jigawa, and Oyo) while also evaluating sustainment of hypertension control in the Federal Capital Territory.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old),
* Elevated blood pressure (SBP ≥ 140 mmHg or DBP ≥ 90 mmHg) documented or measured by a health care professional (e.g., physician, community health extension worker, or community health officer) on two separate occasions or taking a BP-lowering medication, or a history of hypertension.
* Pregnant women are eligible for this program, or
* Cognitively impaired adults are eligible for this program..

Exclusion Criteria:

This program will not include any of the following special populations:

* Individuals who are not yet adults (minors): i.e. infants, children, or teenagers <18 years old, or
* Prisoners or other detained individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Outcome | 36 months
  Difference in the 6-month rolling average of hypertension control between the pre-implementation and implementation periods (defined as <140/<90 mm Hg)
Primary Implementation Outcome | 36 months
  Dose of quarterly supportive supervision visits measured by the proportion of observed/expected visits during the implementation period.

SECONDARY OUTCOMES:
Secondary Effectiveness outcome (hypertension treatment) | 36 months
  Difference in hypertension treatment in the 6-month rolling average between the pre-implementation and implementation periods
Secondary Effectiveness Outcomes (mean systolic blood presure) | 36 months
  Difference in mean systolic blood pressure in the 6-month rolling average between the pre-implementation and implementation periods
Secondary Effectiveness Outcome (mean diastolic blood pressure) | 36 months
  Difference in mean diastolic blood pressure in the 6-month rolling average between the pre-implementation and implementation periods
Secondary Implementation Outcomes: Proportion of selected PHCs who participated in baseline hypertension training | 36 months
  A = Number of PHCs who participated in baseline hypertension training B = Total number of selected PHCs
  Calculation: A ÷ B
Secondary Implementation Outcome: Proportion of selected PHCs who participated in site initiation training | 36 months
  A = Number of PHCs who participated in site initiation training B = Total number of selected PHCs
  Calculation: A ÷ B
Secondary Implementation Outcome: Proportion of selected PHCs who received at least one supportive supervision visit in the past 12 months | 36 months
  A = Number of PHCs who received at least one supportive supervision visit in the past 12 months B = Total number of selected PHCs
  Calculation: A ÷ B
Secondary Implementation Outcome: Proportion of selected PHCs who received an audit and feedback report within the past 3-months | 36 months
  A = Number of PHCs who received at least an audit and feedback report within the past 3-months B = Total number of selected PHCs
  Calculation: A ÷ B
Secondary Implementation Outcome: Percentage of PHCs with a working blood pressure monitor at the site on the day of assessment | 36 months
  A = Number of PHCs with a working blood pressure monitor at the site on the day of assessment (time point: last supervision visit) B = Total number of selected PHCs
  Calculation: A ÷ B
Secondary Implementation Outcome: Percentage of PHCs with blood pressure medicines available on the day of assessment | 36 months
  A = Number of PHCs with blood pressure medicines available on the day of assessment (time point: last supervision visit) B = Total number of selected PHCs
  Calculation: A ÷ B
Secondary Implementation Outcome: Percentage of patients with step up indicated who received step up treatment in the last 6-months | 36 months
  A = Number of patients who need step up treatment and received it
  B = Total number of patients who are registered per month
  Calculation: A ÷ B, 6-monthly rolling average rate
Secondary Implementation Outcome: Number and proportion of adult patients with hypertension who are registered/total number of adult patients with elevated blood pressure within participating PHCs within the past 3 working days | 36 months
  A = Total number of adult patients who had high BP visits to the health facility within the given dates
  B = Total number of patients visits to the health facility within the given dates
  Calculation: A ÷ B
Secondary implementation Outcome: Monthly proportion of registered patients with appropriate stepped care/total number of registered patients | 36 months
  A = Number of patients who need step up treatment and received it
  B = Total number of patients who are registered per month
  Calculation: A ÷ B, 6-monthly rolling average rate
Secondary Implementation Outcome: Monthly proportion of registered patients treated with fixed dose combination therapy/total number of patients on treatment | 36 months
  A = Number of patients who are treated with fixed dose combination therapy
  B = Total number of patients who are treated per month
  Calculation: A ÷ B, 6-month rolling average rate

OTHER OUTCOMES:
Safety Outcome: between-period (pre-implementation versus implementation) differences in the proportion of serious adverse events | 36 months
  Safety Outcome: between-period (pre-implementation versus implementation) differences in the proportion of serious adverse events
Safety Outcome: between-period (pre-implementation versus implementation) differences in the proportion of adverse events of special interest | 36 months
  i.e., clinically ascertained angioedema, syncope, lightheadedness/dizziness, edema, inappropriate medication prescription [e.g., ACE or ARB among patients who are pregnant]
Safety Outcome: Between-period (pre-implementation versus implementation) differences in the proportion of hyperkalemia, hypokalemia, and acute kidney injury | 36 months
  Hyperkalemia, hypokalemia, and acute kidney injury measured in a subset of 5 sites and 250 patients (n=500 total) in both pre-implementation and implementation periods.

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared through NHLBI BioData Catalyst
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 1 year of study conclusion
Access Criteria: Access to study data will be managed through NHLBI BioData Catalyst.

DOCUMENTS (1):
  • Study Protocol (2026-01-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT07351162/Prot_000.pdf